CLINICAL TRIAL: NCT03614585
Title: Exercise Intensity Matters: An Opportunity to Promote Neurorecovery and Cardiovascular Health in Stroke
Brief Title: Exercise Intensity Matters in Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: McMaster University (Other); Jewish Rehabilitation Hospital (Other); Ontario Stroke Network (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marc Roig, Assistant Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 388320
Record Dates: First submitted 2018-07-26; First posted 2018-08-03 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Neurosciences; Exercise; Neurorecovery; Cardiovascular health; High-intensity interval training; Moderate-intensity continuous training
MeSH Terms: conditions — Stroke; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Intensity will be determined using a combination of heart rate reserve (HRR, calculated as HRR= [max HR - resting HR] x [% training] + [resting HR]) and ratings of perceived exertion (RPE). The protocol will involve 10 60-second intervals of high intensity interspersed with 9 60-second low-intensity intervals. The initial high intensity intervals will start at 80% of the HRR (RPE=14-17) and progress by 10% every 4 weeks. Low intensity intervals will be performed at 30% of HRR (RPE=9-11). Three-minute warm-up and 2-minute cool-down periods will be performed at 30% of HRR. Total HIIT time including warm-up and cool-down is 24 minutes.
  Interventions: Behavioral: 12 weeks of High-intensity Interval Training
- Moderate-intensity continuous training (Experimental): Intensity will be determined using a combination of heart rate reserve (HRR, calculated as HRR= [max HR - resting HR] x [% training] + [resting HR]) and ratings of perceived exertion (RPE). The MICT protocol will be increased using a progression schedule previously used (initial intensity at 40% HRR (RPE=9-11), and progressed by 10% HRR every 4 weeks up to 60% HRR (RPE=13-14) will be maintained until the end of the intervention). A 3-minute warm-up and 2-minute cool-down will be performed at 30% HRR (RPE=9-11). The total duration of MICT, including warm-up and cool-down, will be 35 minutes.
  Interventions: Behavioral: 12 weeks of Moderate-Intensity Continuous Training

INTERVENTIONS:
Behavioral: 12 weeks of High-intensity Interval Training — Cardiovascular exercise
  Arms: High-intensity interval training
Behavioral: 12 weeks of Moderate-Intensity Continuous Training — Cardiovascular exercise
  Arms: Moderate-intensity continuous training

SUMMARY:
The main objective of this multi-site project is to compare the effects of 12 weeks of HIIT vs. MICT on brain plasticity. The effects of HIIT vs. MICT on cardiovascular health, psychosocial predictors of physical activity and motor function will also be compared. HIIT and MICT will be delivered through a whole-body exercise paradigm using a recumbent stepper that requires arm and leg forces. Outcomes will be assessed at baseline (T0, 0 weeks), at the end of the intervention (T1, 12 weeks) and at 8-week follow-up (T2, 20 weeks).

DETAILED DESCRIPTION:
Background: Stroke is a major health issue in Canada, with 405,000 Canadians currently living with stroke. Exercise is an important component of stroke rehabilitation that can result in improved function and health. Traditionally, exercise rehabilitation programs for stroke employ moderate-intensity continuous training (MICT) protocols that are typically sustained for 20-30 minutes. The continuous nature of this form of training however, even at moderate intensities, is challenging for many individuals with stroke to sustain due to neuromotor impairments and poor exercise capacity. High-intensity exercise, when delivered in short interval bursts (i.e. high-intensity interval training, HIIT), may be a feasible alternative that allows higher intensities to be achieved during exercise. This is important because intensity of training is the critical factor in promoting changes in neuroplasticity and cardiovascular health, the two most important aspects of recovery and secondary prevention after stroke. Interventions implemented earlier following stroke are generally viewed to yield greater benefits, but high intensity exercise may also promote neuroplasticity and optimize cardiovascular health in later stages of recovery. Furthermore, determining if HIIT is viewed to be motivating and enjoyable for individuals post-stroke can provide insight into the sustainability of this intervention.

Objective: To compare the effects of 12 weeks of HIIT and MICT on neuroplasticity, cardiovascular health and psychosocial predictors of physical activity in individuals with chronic stroke.

Design: Participants will be recruited from two research sites and randomly allocated into HIIT or MICT. Participants will be assessed before and after the training period, and at an 8-week follow-up.

Outcomes: 1) The investigators will assess: Neuroplasticity: by measuring markers of corticospinal excitability at rest and in response to a non-invasive brain stimulation protocol applied over the primary motor cortex (M1); 2) Cardiovascular health: by measuring cardiorespiratory fitness, resting blood pressure, arterial stiffness, and waist-hip ratio; 3) Psychosocial predictors of physical activity: by measuring exercise motivation and enjoyment.

Methods: Neuroplasticity: motor evoked potentials amplitude, intracortical facilitation and short-intracortical inhibition on the lesioned and unlesioned upper limb M1 area at rest and in response to continuous theta-burst will be measured with transcranial magnetic stimulation; Cardiovascular health: cardiorespiratory fitness will be measured with a graded exercise test, resting blood pressure with an automated blood pressure monitor and arterial stiffness using applanation tonometry. Exercise motivation and enjoyment will be assessed with the Physical Activity Enjoyment Scale and the Behavioral Regulation Exercise Questionnaire-3, respectively.

Expected results: Both HIIT and MICT will result in improvements in outcomes of neuroplasticity and cardiovascular health. However, improvements with HIIT will be greater and will last longer. Participants will rate HIIT as enjoyable as MICT, and motivation for exercise will increase similarly after both interventions.

Impact: HIIT is a promising, time-efficient, and potentially more effective alternative to traditional MICT protocols that could offer an opportunity for greater improvement in motor recovery and cardiovascular health in people living with stroke.

ELIGIBILITY:
Inclusion Criteria:

* 6-60 months following first-ever, single stroke confirmed by MRI/CT
* Living in the community and able to independently walk at least 10 meters (assistive devices permitted, as this is representative of many people who regain some walking ability following stroke but commonly with some adaptation)
* Montreal Cognitive Assessment score >20 (individuals with this score are capable to follow exercise instructions)

Exclusion Criteria:

* Significant disability as determined by modified Rankin scale score <2
* Stroke of non-cardiogenic origin or tumor
* Actively engaged in stroke rehabilitation services or a structured exercise program besides the one provided in the study
* Class C or D American Heart Association Risk Criteria
* Other neurological or musculoskeletal co-morbidities that preclude exercise participation
* Pain which is worsened with exercise
* Cognitive, communication, or behavioral issues that would limit safe exercise participation
* Contraindications to transcranial magnetic stimulation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cortico-spinal excitability | 12 weeks
  Single pulse of transcranial magnetic stimulation protocol.

SECONDARY OUTCOMES:
Intra-cortical inhibition | 12 weeks
  Paired-pulse of transcranial magnetic stimulation protocol.
Intra-cortical facilitation | 12 weeks
  Paired-pulse of transcranial magnetic stimulation protocol.
Systolic resting blood pressure | 12 weeks
  Supine resting blood pressure.
Diastolic resting blood pressure | 12 weeks
  Supine resting blood pressure.
Arterial stiffness | 12 weeks
  Central pulse wave velocity.
Cardiorespiratory fitness | 12 weeks
  Maximum rate of oxygen consumption measured during maximum physical effort.
Waist-hip ratio | 12 weeks
  Ratio of waist circumference measured at the level of the umbilicus, and hip circumference taken at the level of the greater trochanters.

OTHER OUTCOMES:
Enjoyment | 12 weeks
  The Physical Activity Enjoyment Scale. Each item is scored 1-7 (1=does not make me happy, 7=makes me happy), yielding a total between 8 and 56.
Motivation | 12 weeks
  The Behavioral Regulation Exercise Questionnaire-3. 24 items using a 5-point Likert scale (0=Not true for me, 4=Very true for me).
Gait speed | 12 weeks
  self- and fast-paced 6-meter gait speed.
Walking capacity | 12 weeks
  6-Minute Walk Test.
Motor learning | 12 weeks
  A motor task that requires modulating hand-grasping force. The goal is to apply force, move the cursor, and reach targets displayed on the screen as accurately as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Roig, PhD, Principal Investigator — McGill University; Ada Tang, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Ontario Central South Stroke Network, Hamilton, Ontario
  - Jewish Rehabiliation Hospital, Laval, Quebec

IPD SHARING:
Plan to Share IPD: No
Results will be publish in peer-review journals.

REFERENCES:
- [Derived] Rodrigues L, Moncion K, Angelopoulos SA, Heras BL, Sweet S, Eng JJ, Fung J, MacKay-Lyons M, Tang A, Roig M. Psychosocial Responses to a Cardiovascular Exercise Randomized Controlled Trial: Does Intensity Matter for Individuals Post-stroke? Arch Phys Med Rehabil. 2025 Jun;106(6):828-836. doi: 10.1016/j.apmr.2025.01.468. Epub 2025 Jan 31. PMID 39894292
- [Derived] Moncion K, Rodrigues L, De Las Heras B, Noguchi KS, Wiley E, Eng JJ, MacKay-Lyons M, Sweet SN, Thiel A, Fung J, Stratford P, Richardson JA, MacDonald MJ, Roig M, Tang A. Cardiorespiratory Fitness Benefits of High-Intensity Interval Training After Stroke: A Randomized Controlled Trial. Stroke. 2024 Sep;55(9):2202-2211. doi: 10.1161/STROKEAHA.124.046564. Epub 2024 Aug 7. PMID 39113181
- [Derived] Rodrigues L, Moncion K, Eng JJ, Noguchi KS, Wiley E, de Las Heras B, Sweet SN, Fung J, MacKay-Lyons M, Nelson AJ, Medeiros D, Crozier J, Thiel A, Tang A, Roig M. Intensity matters: protocol for a randomized controlled trial exercise intervention for individuals with chronic stroke. Trials. 2022 May 24;23(1):442. doi: 10.1186/s13063-022-06359-w. PMID 35610659